CLINICAL TRIAL: NCT01756053
Title: A Pilot Feasibility Study of the Effects of ABT-089 on Smoking Abstinence Symptoms and Reward
Brief Title: Effects of ABT-089 on Smoking Abstinence Symptoms and Reward
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial discontinued based on the results of an interim futility analysis.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 815238
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-02

CONDITIONS: Nicotine Addiction
Keywords: Smoking; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — pozanicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-089 (Active Comparator): During both 10-day study medication periods (Days 1-10 & Days 32-41), subjects will take 4 capsules daily. Administration of study medication will be double-blind and in counter-balanced order.
  Those randomized to active ABT-089 during study medication period 1 will take four 10mg capsules daily (40mg daily) during the 10-day medication period. During study medication period 2, these subjects will take four capsules of the matched placebo capsules.
  Interventions: Drug: ABT-089
- Placebo (Placebo Comparator): These are matched placebo capsules manufactured by the study drug supplier.
  During both 10-day study medication periods (Days 1-10 & Days 32-41), subjects will take 4 capsules daily. Administration of study medication will be double-blind and in counter-balanced order.
  Those randomized to matched placebo during study medication period 1 will take four capsules daily during the 10-day medication period. During study medication period 2, these subjects will take four 10mg capsules (40mg daily) of the active ABT-089 capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-089 — Selective neuronal nicotinic receptor agonist.
  Other Names: Pozanicline
  Arms: ABT-089
Drug: Placebo — Matched placebo capsules supplied by study drug supplier.
  Arms: Placebo

SUMMARY:
This Phase IIa within-subject, cross-over pilot study will evaluate the effects of ABT-089 (an experimental medication not approved by the FDA) when administered as 40mg oral once daily dose for 10 days, compared to placebo, on the following: abstinence-induced cognitive deficits, smoking withdrawal, smoking urges, smoking reward, and a brief, monitored quit attempt (~4 days). The key cognitive domains include: working memory, sustained attention, and response inhibition.

DETAILED DESCRIPTION:
This is a single-site, phase IIa, double-blind, within-subject, cross-over, human laboratory study. Subjects will be healthy, treatment-seeking female and male adult smokers, ages 18 to 65 years old. Subjects deemed eligible for participation after an Intake Visit (~Day -7) will complete baseline assessments and receive period 1 medication (ABT-089 or placebo) at the Baseline Visit (Day 0). Subjects will take 40mg of ABT-089 or placebo, based on random assignment, every day for two identical 10-day study treatment periods.

Subjects will begin period 1 study medication on Day 1. On Days 3 and 5, subjects will complete in-clinic medication run-up and monitoring assessments. On Day 5, subjects will begin a ~24-hour period of mandatory abstinence from smoking. Day 6 is conducted in two parts. Part 1 will consist of confirmation of smoking abstinence, testing for abstinence-induced cognitive deficits and the collection of subjective assessments. Part 2 will begin with a programmed smoking lapse, after which the subjective rewarding value of the programmed lapse cigarette will be assessed. Before leaving the clinic on Day 6, subjects will receive brief cessation counseling and be instructed to try to remain abstinent from 10pm that evening until after the final Observation Visit on Day 10.

During the ~4-day monitored abstinence/observation phase, subjects will complete in-clinic observation visits (subjective assessments, medication adherence, etc.) on Days 7, 8, and 10.

After a ~3-week medication washout period and Period 2 Medication Pick-up Visit on ~Day 31, subjects will begin study medication (either ABT-089 or placebo; but will always be the opposite of the assigned study medication in period 1) and participate in period 2 of the study following the same procedures as period 1.

ELIGIBILITY:
Inclusion Criteria.

Eligible subjects will be:

1. Male and female smokers who are between 18 and 65 years of age and self-report smoking at least 10 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months.
2. Healthy as determined by the Study Physician, based on relevant medical history, physical examination (including vitals), and basic screening tests (CBC, CHEM7, AST/ALT).
3. Smokers who wish to quit smoking in the next 2-6 months (treatment-seeking), because our prior work suggests that motivated subjects are more sensitive to medication effects on smoking behavior. Using a scale from 0 to 100 (100, being extremely interested), subjects must rate their interest in quitting smoking within the next 6 months greater than 50.
4. Able to communicate fluently in English (speaking, writing, and reading).
5. Plan to live in the area for the next 2 months.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Exclusion Criteria.

Subjects who self-report and/or present with the following criteria will not be eligible to participate in the study:

1. Smoking behavior.

   1. Current enrollment or firm plans to quit smoking and/or enroll in a smoking cessation program within the next 2 months.
   2. Current and/or anticipated use of any nicotine substitutes and/or smoking cessation treatments/medications within the next 2 months.
   3. Provide a Carbon Monoxide (CO) reading less than 11 parts per million (ppm) at Intake.
   4. Provide a CO reading of 10 ppm or greater at either Testing Visit (Days 6 and 37). If the CO reading is greater than or equal to 10 ppm, but there is a 50% reduction from the CO reading collected at the Baseline/Period 1 Medication Pick-Up Visit, this will be sufficient and the subject may continue as scheduled.
   5. Self-report smoking during the mandatory abstinence period at either Testing Visit (Days 6 and 37).
   6. Regular use of chewing tobacco or snus.
2. Alcohol/Drugs.

   1. History of substance abuse in the past 6 months and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana, or stimulants). Subjects reporting a history of substance abuse must be in remission at least 6 months or greater.
   2. Current alcohol consumption that exceeds 25 standard drinks/week.
   3. Provide a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 at Intake, Baseline/Period 1 Medication Pick-Up, or Testing Visits (Days 6 and 37).
   4. A positive urine drug screen for cocaine, PCP, amphetamines, methamphetamines, tricyclic antidepressants, opiates, methadone, benzodiazepines, and/or barbiturates at Intake, Baseline/Period 1 Medication Pick-Up, Period 2 Medication Pick-Up, and Observation Visits on Days 10 and 41.
3. Medical.

   1. Women who are pregnant, planning a pregnancy, and/or breast feeding. All female subjects will undergo a urine pregnancy test at Intake, after which only females determined to be of childbearing potential will complete a urine pregnancy test at Baseline/Period 1 Medication Pick-Up, Period 2 Medication Pick-Up, and Observation Visits on Days 10 and 41. By signing the combined consent and HIPAA form, women of childbearing potential agree to use an approved method of contraception during the study.
   2. Men who do not agree to use an approved method of contraception during the study. Men who are sexually active must be surgically sterile (vasectomy) or using a barrier method (condom) of birth control for the duration of the study. By signing the combined consent and HIPAA form, men agree to use an approved method of contraception.
   3. Current treatment of cancer or diagnosed with cancer (except basal cell carcinoma) in the past 6 months.
   4. Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing neurocognitive task performance.
   5. Color blindness.
   6. History of brain injury.
   7. History of epilepsy or a seizure disorder.
   8. Low or borderline intellectual functioning - determined by receiving a score of less than 90 on the Shipley Institute of Living Scale (SILS, administered at Intake), which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test.
   9. Serious or unstable disease within the past 6 months (i.e., heart disease, liver/kidney failure).
   10. Recent history (last 6 months) of abnormal heart rhythms, tachycardia, and/or cardiovascular disease (stroke, angina, heart attack) may result in ineligibility. These conditions will be evaluated on a case-by-case basis by the Study Physician.
   11. Clinically significant abnormalities determined by physical examination and collection of vital signs at Intake. Abnormalities will be assessed by the Study Physician and eligibility will be determined on a case-by-case basis.
   12. Uncontrolled hypertension (Systolic Blood Pressure [SBP] greater than or equal to 160 mmHg and/or Diastolic Blood Pressure [DBP] greater than or equal to 100 mmHg).
   13. Heart rate/pulse greater than or equal to 110 beats per minute (bpm).
   14. Clinically significant abnormalities in clinical chemistry (CBC, CHEM7, and AST/ALT). Results greater than 20% outside of normal range will be evaluated for clinical significance by the Study Physician and eligibility will be determined on a case-by-case basis.
   15. Inability to provide an assessable blood sample for basic screening tests (CBC, CHEM7, and AST/ALT) at Intake.
4. Psychiatric.

   As determined by self-report, the Mini International Neuropsychiatric Interview (MINI), and/or Columbia-Suicide Severity Rating Scale (C-SSRS):
   1. Any suicide risk score on the MINI.
   2. Current (past month) suicidal ideation or lifetime suicidal behavior on the C-SSRS.
   3. Lifetime history or current diagnosis of psychosis, bipolar disorder, and/or schizophrenia.
   4. Current diagnosis of major depression and/or recurrent major depression. Persons with a history of a single episode of major depression, in remission for 6 months or longer, are eligible provided they are not excluded based on medications (see Medication Exclusion Criteria).
   5. Current or past hypomanic/manic episode.
   6. History or current diagnosis of posttraumatic stress disorder (PTSD).
   7. Prior or current diagnosis of attention deficit hyperactivity disorder (ADHD).
5. Medication.

   1. Current use or recent discontinuation (within the last 14 days at the time of Intake) of:

      * Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix).
      * Anti-anxiety or panic disorder medications.
      * Anti-psychotic medications.
      * Medications used to treat depression (e.g., Wellbutrin, MAOIs, SSRIS, tricyclic antidepressants).
      * Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
      * Systemic corticosteroids.
   2. Current use of:

      * Nicotine replacement therapy (NRT).
   3. Daily use of:

      * Opiate-containing medications for chronic pain.
      * Inhaled corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: CIRNA Center homepage — http://www.med.upenn.edu/cirna/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty three subjects were consented and screened for eligibility at an Intake Visit between April 2013 and December 2013 at the Center for Interdisciplinary Research on Nicotine Addiction (Philadelphia, PA).
Pre-assignment Details: Seventeen of the 53 subjects were randomized and received study medication. Of those NOT randomized, 30 were deemed ineligible and 6 withdrew from the study.
Groups:
- ABT-089, Then Placebo: Those randomized to active ABT-089 during study medication period 1 will take four 10mg capsules daily (40mg daily) during a 10-day medication period. After a washout period of ~21 days, these subjects will then take four capsules of matching placebo daily for a second 10-day medication period.
  ABT-089: Selective neuronal nicotinic receptor agonist.
- Placebo, Then ABT-089: Those randomized to placebo (matching ABT-089 10 mg capsules) during study medication period 1 will take four capsules daily during a 10-day medication period. After a washout period of ~21 days, these subjects will then take four 10 mg capsules (40 mg) daily of ABT-089 for a second 10-day study medication period.
  Placebo: Matching placebo capsules supplied by study drug supplier.
Period: Period 1 (10 Days)
Arm/Group | ABT-089, Then Placebo | Placebo, Then ABT-089
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Washout Period (~21 Days)
Arm/Group | ABT-089, Then Placebo | Placebo, Then ABT-089
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Period 2 (10 Days)
Arm/Group | ABT-089, Then Placebo | Placebo, Then ABT-089
Started | 7 | 8
Completed | 7 | 6
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Subjects: Subjects who were randomized and received their Period 1 study medication (ABT-089 or matching placebo).
Arm/Group | All Study Subjects
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.76471 (11.20563)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Abstinence-induced Cognitive Deficits (N-Back Accuracy)
Description: We will assess whether ABT-089 ameliorates the cognitive deficits due to smoking abstinence.
  To assess, all subjects will complete a computerized N-Back task during the Testing Day Session (Days 6 & 37) in each study medication period. Each Testing Day session occurs after 24 hours of abstinence from smoking. During one study medication period, subjects will take active ABT-089; during the other period, subjects will take a matched placebo.
  Each of the task conditions (0-, 1-, 2-, and 3-back) will be administered in a pseudorandomized counterbalanced order. Each difficulty level will consist of one block of 50 trials, preceded by a practice block of 20 trials. The primary dependent variables for this task are total number of correct responses (out of 60) and reaction time (milliseconds).
  All computerized neurocognitive tasks are completed in a quiet, standardized environment in our clinic.
  NOTE: Each PPT completes 1 Baseline (no tx.) and 2 Testing Days (ABT/Placebo)
Time Frame: Baseline (Day 0) and Test Day (Days 6 & 37)
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Number of correct responses (out of 60)
Groups:
- ABT-089: Subjects who were assigned to active ABT-089 (four 10 mg capsules daily) in either Period 1 or Period 2 of the study. Each study period is 10 days.
- Placebo: Subjects who were assigned to matched placebo (four capsules daily) in either Period 1 or Period 2 of the study. Each study period is 10 days.
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Number of correct responses (out of 60)
  Baseline (Day 0) | 44.2 (7.2) | 44.2 (7.2)
  Test Days (Days 6 & 37) | 47.5 (8.4) | 47.5 (8.4)

2. Secondary Outcome: Effects of ABT-089 on Mood
Description: PANAS: The Positive and Negative Affect Schedule (PANAS), a 20-item Likert-format self-report measure, was used to assess Positive Affect (PA; 10 items, e.g., enthusiastic, strong) and Negative Affect (NA; 10 items, e.g., distressed, upset), two dominant and generally orthogonal dimensions of affect. Scores for the 10 items on each subscale were summed to create summary scores (range: 10-50); higher scores indicate greater intensity of mood (i.e., more positive or more negative affect). Higher ratings of positive affect and lower ratings of negative affect are considered better outcomes.
Time Frame: Days 6 and 37
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Scores on a scale
  PANAS: Positive Affect | 25.4 (9.2) | 26.2 (9.6)
  PANAS: Negative Affect | 13.2 (3.6) | 13.5 (4.6)

3. Secondary Outcome: Effects of ABT-089 on Withdrawal Symptoms
Description: MNWS: The Minnesota Nicotine Withdrawal Scale - Revised version captures the current state of nicotine withdrawal. The scale assesses 15 items of nicotine withdrawal (including 7 DSM-IV items) such as: dysphoria or depressed mood, insomnia, irritability/frustration/anger, anxiety, difficulty concentrating, restlessness, and increased appetite/weight gain. Subjects will rate the intensity of their symptoms on the following scale: 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe. A "withdrawal discomfort score" was calculated as the sum of the first 9 items (possible range: 0-36) and is a well-validated measure of nicotine withdrawal; a higher score indicates more severe withdrawal.
Time Frame: Days 6 and 37
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Scores on a scale | 6.8 (6.1) | 6.6 (6.7)

4. Secondary Outcome: Effects of ABT-089 on Smoking Urges/Craving
Description: QSU-B: The 10-item brief QSU (QSU-B) questionnaire was used to assess smoking urges. Each item is rated on a 7-point scale (1 = strongly disagree, 7 = strongly agree). A total score is calculated as the sum of the individual items (range: 10-70). Higher scores indicate more severe urges to smoke.
Time Frame: Days 6 and 37
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Scores on a scale | 37.4 (17.2) | 38.3 (15.8)

5. Secondary Outcome: Effects of ABT-089 on Attention-deficit and Hyperactive Symptoms
Description: ADHD symptoms: The 27-item BAARS-IV scale was used to assess current attention-deficit and hyperactive symptoms. Participant rated the intensity of their symptoms using the following scale: 1= never or rarely, 2 = sometimes, 3 = often, or 4 = very often. A total score was calculated as the sum of the individual items (range: 27-108). Higher scores indicate more frequent ADHD symptoms.
Time Frame: Days 6 and 37
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Scores on a scale | 33.2 (6.8) | 35.4 (9.6)

6. Secondary Outcome: Effects of ABT-089 on Cigarette Ratings
Description: Cigarette evaluation scale: The Cigarette Evaluation Scale (CES), developed to assess subjective effects of smoking, is an 11-item Likert-format measure. Questions include items for nausea and dizziness, craving relief, and enjoyment of airway sensations. Items are rated on a scale from 1 ("Not at all") to 7 ("Extremely); a summary score is calculated as the mean of all responses (range: 1-7). Higher scores indicate stronger subjective effects of smoking.
Time Frame: Days 6 and 37
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Scores on a scale | 2.8 (0.78) | 2.9 (0.76)

7. Secondary Outcome: Effects of ABT-089 on Days of Biochemically-confirmed Abstinence
Description: Daily smoking rate will be assessed at each in-person visit using the Timeline Follow-Back assessment. Abstinence will be confirmed by exhaled carbon monoxide levels during a ~4-day monitored abstinence phase within each period.
Time Frame: Days 7, 8, 9, 10, 38, 39, 40, & 41
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Days of abstinence
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Days of abstinence | 1.2 (1.7) | 1.2 (1.8)

8. Primary Outcome: Change in Abstinence-induced Cognitive Deficits (N-Back Correct Response Time)
Description: as for outcome 1
Time Frame: Baseline (Day 0) and Test Day (Days 6 & 37)
Population: Only participants completing both study periods (n=13) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | ABT-089 | Placebo
Number analyzed (Participants) | 13 | 13
Milliseconds
  Baseline (Day 0) | 612.4 (125.5) | 612.4 (125.5)
  Test Days (Days 6 & 37) | 646.5 (143.3) | 638.9 (129.5)

ADVERSE EVENTS:
Time Frame: 10 days for each study medication period (ABT-089/Placebo in counter-balanced order)
Description: The safety population described within this section includes all subjects who received at least one dose of ABT-089 (n=16) or Placebo (n=16).
  Systematic Assessment: Subjects completed a side effect checklist at every in-person study visit over the course of the treatment period. Subjects could also spontaneously report AEs at any time.
Groups:
- ABT-089: Subjects were assigned to take four 10 mg capsules daily (40 mg daily) during a 10-day medication period.
  ABT-089: Selective neuronal nicotinic receptor agonist.
- Placebo: Subjects were assigned to take four placebo capsules (matching ABT-089 10 mg) daily during a 10-day medication period.
  Placebo: Matched placebo capsules supplied by study drug supplier.
Arm/Group | ABT-089 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-089 (N=16) | Placebo (N=16)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (4)
Fatigue (General disorders) | 2 (3) | 3 (4)
Irritability (General disorders) | 8 (22) | 11 (30)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2)
Headache (Nervous system disorders) | 2 (7) | 6 (12)
Anxiety (Psychiatric disorders) | 6 (18) | 8 (20)
Hostility (Psychiatric disorders) | 3 (7) | 7 (17)
Tension (Psychiatric disorders) | 5 (16) | 7 (21)
Depressed Mood (Psychiatric disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 9 (20) | 9 (21)
Vivid Dreams (Psychiatric disorders) | 4 (4) | 4 (6)
Insomnia (Psychiatric disorders) | 2 (6) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) — Runny Nose
Pyrexia (General disorders) | 1 (1) | 0 (0) — Fever
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) — Sore Throat
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Muscle pain

LIMITATIONS AND CAVEATS:
The study was terminated early due to the results of an interim futility analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes